CLINICAL TRIAL: NCT06728215
Title: CRET Therapy in Low Back Pain Treatment.
Brief Title: Capacitive-Resistive Energy Transfer (CRET) for the Treatment of Low Back Pain
Status: Completed | Type: Observational
Sponsor: D&V FARMA srl (Industry)
Responsible Party: Sponsor
Other Study IDs: FISIO01
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- UNIQ capacitive/resistive electrode: subjects with LBP treated with Fisiowarm 7.0 and the new capacitive/resistive electrode (UNIQ electrode Fisiowarm 7.0, Golden Star Srl, Rome, Italy), for 15' at a frequency of 300 KHz (Treated Group)
  Interventions: Device: CRET 1
- monopolar electrode group: Subject with LBP treated with a classical methodology using the monopolar electrode Activ CT8 INDIBA® at a frequency of 448 KHz in both resistive and capacitive modes, for 10 min each mode with two different electrodes. (Control group).
  Interventions: Device: CRET 2

INTERVENTIONS:
Device: CRET 1 — Fisiowarm 7.0 and the new capacitive/resistive electrode, for 15' at a frequency of 300 KHz (Treated Group).
  Groups: UNIQ capacitive/resistive electrode
Device: CRET 2 — Classical methodology using the monopolar electrode Activ CT8 INDIBA® at a frequency of 448 KHz in both resistive and capacitive modes, for 10 min each mode with two different electrodes. (Control group).
  Groups: monopolar electrode group

SUMMARY:
This retrospective observational study compares the effectiveness of two CRET therapies in adults with physical dysfunction. It evaluates whether the UNIQ electrode Fisiowarm 7.0 improves lumbar ROM (Schober test) and reduces pain (VAS scores) more effectively than the classical methodology, with assessments at baseline (T0) and two weeks (T1).

DETAILED DESCRIPTION:
The goal of this retrospective observational study is to compare the effectiveness of two CRET therapy methodologies in adults (mean age ±SD: 51.23±16.89 for treated, 51.20±14.34 for control; M/F ratio: 42%M, 58%F for treated, 40%M, 60%F for control) experiencing physical dysfunction.

The main questions it aims to answer are:

* Does treatment with the UNIQ electrode Fisiowarm 7.0 improve range of motion (ROM) as measured by the Schober test more effectively than the classical methodology?
* Does treatment with the UNIQ electrode Fisiowarm 7.0 reduce pain levels, as reported through VAS scores, more effectively than the classical methodology?

Participants underwent therapy with either Fisiowarm 7.0 or Activ CT8 INDIBA® as per their group assignment.

Have their ROM measured using the Schober test at baseline (T0) and after two weeks (T1).

Report VAS scores before therapy (T0) and after two weeks (T1) to assess pain levels.

ELIGIBILITY:
Inclusion criteria

* age 18 years old or older
* reported a visual analogic scale (VAS) for pain equal or greater than 6 cm
* a ROM measured by Schober test
* naïve to CRET therapy
* non-concomitant physiotherapy treatment (e.g. diathermy, laser therapy etc..).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data derived from subject affected by low back pain.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
VAS | 2 WEEKS
  The Visual Analog Scale (VAS) measures pain intensity on a scale of 1 to 10, where 1 represents "no pain" and 10 represents "worst imaginable pain."

SECONDARY OUTCOMES:
ROM | 2 WEEKS
  The Schober test measures the range of motion (ROM) in the lumbar spine during forward bending, with a normal increase of 4-7 cm indicating good flexibility. An increase of less than 4 cm suggests restricted lumbar mobility, often associated with spinal disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Alessio Papaianopol, Doctor, Study Director — Ti Riabilita
Locations (1):
- Ars Fisio, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Koes BW, van Tulder MW, Thomas S. Diagnosis and treatment of low back pain. BMJ. 2006 Jun 17;332(7555):1430-4. doi: 10.1136/bmj.332.7555.1430. No abstract available. PMID 16777886
- [Background] Kim GW, Won YH, Park SH, Seo JH, Kim DH, Lee HN, Ko MH. Effects of a Newly Developed Therapeutic Deep Heating Device Using High Frequency in Patients with Shoulder Pain and Disability: A Pilot Study. Pain Res Manag. 2019 May 2;2019:8215371. doi: 10.1155/2019/8215371. eCollection 2019. PMID 31191789
- [Background] Hoy D, Bain C, Williams G, March L, Brooks P, Blyth F, Woolf A, Vos T, Buchbinder R. A systematic review of the global prevalence of low back pain. Arthritis Rheum. 2012 Jun;64(6):2028-37. doi: 10.1002/art.34347. Epub 2012 Jan 9. PMID 22231424
- [Background] Dunabeitia I, Arrieta H, Torres-Unda J, Gil J, Santos-Concejero J, Gil SM, Irazusta J, Bidaurrazaga-Letona I. Effects of a capacitive-resistive electric transfer therapy on physiological and biomechanical parameters in recreational runners: A randomized controlled crossover trial. Phys Ther Sport. 2018 Jul;32:227-234. doi: 10.1016/j.ptsp.2018.05.020. Epub 2018 May 26. PMID 29870922
- [Background] Clijsen R, Leoni D, Schneebeli A, Cescon C, Soldini E, Li L, Barbero M. Does the Application of Tecar Therapy Affect Temperature and Perfusion of Skin and Muscle Microcirculation? A Pilot Feasibility Study on Healthy Subjects. J Altern Complement Med. 2020 Feb;26(2):147-153. doi: 10.1089/acm.2019.0165. Epub 2019 Oct 3. PMID 31580698
- [Background] Chiarotto A, Maxwell LJ, Terwee CB, Wells GA, Tugwell P, Ostelo RW. Roland-Morris Disability Questionnaire and Oswestry Disability Index: Which Has Better Measurement Properties for Measuring Physical Functioning in Nonspecific Low Back Pain? Systematic Review and Meta-Analysis. Phys Ther. 2016 Oct;96(10):1620-1637. doi: 10.2522/ptj.20150420. Epub 2016 Apr 14. PMID 27081203
- [Background] Bardin LD, King P, Maher CG. Diagnostic triage for low back pain: a practical approach for primary care. Med J Aust. 2017 Apr 3;206(6):268-273. doi: 10.5694/mja16.00828. PMID 28359011
- [Background] Barassi G, Mariani C, Supplizi M, Prosperi L, Di Simone E, Marinucci C, Pellegrino R, Guglielmi V, Younes A, Di Iorio A. Capacitive and Resistive Electric Transfer Therapy: A Comparison of Operating Methods in Non-specific Chronic Low Back Pain. Adv Exp Med Biol. 2022;1375:39-46. doi: 10.1007/5584_2021_692. PMID 35147930
- [Background] Bahns C, Happe L, Thiel C, Kopkow C. Physical therapy for patients with low back pain in Germany: a survey of current practice. BMC Musculoskelet Disord. 2021 Jun 19;22(1):563. doi: 10.1186/s12891-021-04422-2. PMID 34147077
- [Background] Amjad F, Mohseni Bandpei MA, Gilani SA, Arooj A. Reliability of modified-modified Schober's test for the assessment of lumbar range of motion. J Pak Med Assoc. 2022 Sep;72(9):1755-1759. doi: 10.47391/JPMA.4071. PMID 36280970